CLINICAL TRIAL: NCT00250757
Title: Prostate Cancer Diagnosis Through NMR Spectroscopy of Semen and Prostatic Secretions
Status: Terminated | Type: Observational
Why Stopped: Study was not renewed timely with IRB of record.
Sponsor: New Mexico Cancer Research Alliance (Other)
Responsible Party: Sponsor
Other Study IDs: 2904C
Record Dates: First submitted 2005-11-04; First posted 2005-11-08 (Estimated); Last update posted 2016-01-08 (Estimated); Status verified 2016-01

CONDITIONS: Prostate Cancer
Keywords: prostate; NMR Spectroscopy
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Semen samples or Prostatic secretions (via prostate massage).
Oversight: Data Monitoring Committee: Yes

SUMMARY:
To develop the hypothesis that quantitative NMR spectroscopy of human semen can be used to diagnose prostate cancer.

DETAILED DESCRIPTION:
Any willing subject who meets the male gender requirements, who is competent, agrees to participate, and is able to understand the consent form.

ELIGIBILITY:
Inclusion Criteria:

* Any willing subject who meets the male gender requirements, who is competent, agrees to participate, and is able to understand the consent form.

Exclusion Criteria:

* Not sepcified.

Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Males with and without Prostate cancer.
Sampling Method: Non-Probability Sample
Enrollment: 101 (Actual)
Dates: Start 2005-10; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Laurel Sillerud, MD, Principal Investigator — University of New Mexico
Locations (1):
- University of New Mexico Cancer Center, Albuquerque, New Mexico, United States